CLINICAL TRIAL: NCT04439474
Title: Determining the Effect of Vitamin D, Dyslipidemia and Microvascular in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Mohammad Sadegh Bagheri Baghdasht, Principal Investigator, Baqiyatallah Medical Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.BMSU.REC.1392.32
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with vitamin D deficiency (Experimental): This group receives 50,000 units of vitamin D3 daily for up to 8 days until the serum level of vitamin D reaches above 30 ng/ml.
  Interventions: Drug: Vitamin D3
- Patients without vitamin D deficiency (Active Comparator): Participants in this group receive only their usual treatments
  Interventions: Drug: Routine treatment

INTERVENTIONS:
Drug: Vitamin D3 — For up to 8 days, 50,000 units of vitamin D3 are given daily to patients in the first group so that the serum level of vitamin D reaches above 30 g / ml.
  Arms: Patients with vitamin D deficiency
Drug: Routine treatment — In this group, patients receive their usual medications and treatments
  Arms: Patients without vitamin D deficiency

SUMMARY:
This study looked at the effect of vitamin D levels on the complications of type 2 diabetes and the fat profile of patients with diabetes.Participants in this study were divided into two groups. One group included participants with vitamin D deficiency and the other group did not.The first group receives 50,000 units of oral vitamin D 3 daily for up to 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Having conscious satisfaction

Exclusion Criteria:

* Patients with a history of gastrointestinal surgery
* Patients with a history of renal failure
* Patients with a history of vitamin D intake and calcium-containing compounds
* Patients with a history of liver disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Vitamin D serum levels | up to 1 year
  Vitamin D serum levels measured by blood tests
Triglyceride | up to 1 year
  Level of blood triglycerides measured by a blood test
Blood cholesterol levels | up to 1 year
  Blood cholesterol levels measured by a blood test
HDL | up to 1 year
  Blood HDL levels measured by a blood test
LDL | up to 1 year
  Blood LDL levels measured by a blood test
Fasting blood glucose | up to 1 year
  Fasting blood glucose levels measured by a blood test
Neuropathy | up to 1 year
  Neuropathy based on United Kingdom Screening TEST
Nephropathy | up to 1 year
  Nephropathy based on albumin excretion evaluation
Retinopathy | up to 1 year
  Retinopathy based on an ophthalmologist's examination
blood pressure | up to 1 year
  Systolic and diastolic blood pressure measured by Sphygmomanometer
HBA1C | up to 1 year
  Blood sugar levels measured in the last three months measured by blood test

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Sadegh Bagheri Baghdasht, Tehran, Iran